CLINICAL TRIAL: NCT00752024
Title: Stereotactic Aspiration and Thrombolysis of Intracerebral Hemorrhage: a Prospective Controlled Study（SATIH）
Brief Title: Stereotactic Aspiration and Thrombolysis of Intracerebral Hemorrhage: a Prospective Controlled Study
Acronym: SATIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Wei Wang and Zhouping Tang, Department of Neurology of Tongji Hospital, Huazhong University of Sci. and Tec.
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006AA301B50-1
Record Dates: First submitted 2008-06-09; First posted 2008-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Hypertensive Intracerebral Hemorrhage
Keywords: HICH; Suction drainages; TTAC
MeSH Terms: conditions — Intracranial Hemorrhage, Hypertensive | interventions — Suction; Hemostasis; Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): To position haematoma's location, drills several millimeter holes in the localization point of puncture, then insert the drainage tube to inhale haematoma, gives the filament resolver interrupted for liquefication drainage afterward.
  Interventions: Device: YL-1 type of intracranial hematoma puncture needle
- 2 (Active Comparator): In the treatment, under the convention we use the dehydrator for patients, the ultra early patient may use anti-filament medicinal preparation 6- amino-caproic acid 6-12g/d, intravenous drip, the period of revolution does not surpass for 24 hours, then just right for the illness treatment.
  Interventions: Drug: dehydrating agent, haemostatic

INTERVENTIONS:
Device: YL-1 type of intracranial hematoma puncture needle — YL-1 type of intracranial hematoma puncture needle(Pat. NO.is ZL：93244252•8) was originated by Beijing WanTeFu Medical Apparatus Co.Ltd in 1997. With integration of needle and bur drill it is designed as hard tunnel.By the technique of skull self-holding, the puncture needle can being fixed in the target of haematoma for several days.This technique is convenient, simple and safe.
  To position haematoma's location, drills 3 millimeter holes in the localization point of puncture, then insert the drainage tube to inhale haematoma, gives the filament resolver interrupted for liquefication drainage afterward.
  Other Names: aspiration drainage
  Arms: 1
Drug: dehydrating agent, haemostatic — In the treatment, under the convention we use the dehydrator for patients, the ultra early patient may use anti-filament medicinal preparation 6- amino-caproic acid 6-12g/d, intravenous drip, the period of revolution does not surpass for 24 hours, then just right for the illness treatment.
  Other Names: conservative treatment
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the superiority of effect of the modified micro-invasive aspiration and drainage and conservative medical therapy in the treatment of ICH spontaneously hypertensive scientifically.

DETAILED DESCRIPTION:
The stereotactic computed tomographic-guided aspiration and drainage is one of the best choices in the treatment of a large-scale deep supratentorial intracerebral hematoma. It uses hardware access technology, in a relatively short time to enter the hematoma center, with suction liquefaction technology. It has the advantage of a higher clearance rate of the hematoma, simple convenience, small trauma and low-cost. We carry on the suitable improvement in this technology's foundation in view of its deficiency, the introduction of the concept of the individual, will further reduce the rate of bleeding and mortality, improve survival, such as long-term quality of life.

We will adopt scales such as the rate of rebleeding, mortality, complication,NIHSS, MRS, BI, GOS scale to analysis and evaluating efficacy and safety of this technology and conservative treatment in the treatment of HICH.

ELIGIBILITY:
Inclusion Criteria:

* CT diagnosis of spontaneous supratentorial intracerebral hemorrhage, the amount of bleeding more than 50 ml, and had neurological signs
* All income groups the incidence of medical records to be random, the time should be < 69 hours to ensure that within 72 hours of the onset of the operation
* To be random, former GCS score > = 5 points
* Systolic blood pressure <= 200 mmHg, mean arterial pressure <= 150 mmHg (if higher than this value, but as corresponding to this standard can be dealt with the group, and only reached the standard before they can ask for random)
* Fasting plasma glucose <= 11.1 mmol / L (if higher than this value, but as corresponding to this standard can be dealt with the group, and only reached the standard before they can ask for random)
* Patients aged 18 to 80-year-old.
* Based on China's relevant laws, the patient himself or family members (only in patients with the loss of his ability to judge the acts of circumstances) agreed to participate in this study, a good compliance, to fully comply with random, in accordance with the decision by the treatment, patients himself Or family members must sign informed consent moreover.
* Patients themselves or their families (only in patients with the loss of his ability to judge the acts of circumstances) have willingness and ability to follow the research program, data collection and preservation of history and follow-up process of informed consent.

Exclusion Criteria:

* Patients clotting mechanisms are obstacles or having the experience of the use of anticoagulant drug (PT> 15s, APTT> 40s, INR> 1.4, platelet count <100 × 10 9 / L).
* Cerebral hernia formed more than two hours
* The merger of other serious system failure (heart, liver and kidney, etc.) or a variety of end-stage disease with cerebral hematoma (such as renal failure late cerebral hemorrhage, blood disease with cerebral hemorrhage)
* Prior to the onset of a variety of reasons for the defect or neurological movement disorder
* A clear cause of cerebral hemorrhage such as intracranial aneurysm, or dynamic
* such as a venous malformation
* Intracranial or serious systemic infection
* Marked cognitive impairment or mental abnormality
* Other such as pregnancy, cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The rate of rebleeding and mortality, Glasgow Outcome Scale for prognosis | duration of 14 days after operation(rebleeding), duration of hospital stay(mortality), 180 days after onset(mortality and GOS)

SECONDARY OUTCOMES:
Nation of Health Stroke Scale Score , modified Rankin Scale, Barthel Index complications | the moment of admission and post operation(NIHSS), 14 days after admission(NIHSS,MRS), duration of hospital stay(complications), 180 days after onset(BI, MRS)

CONTACTS AND LOCATIONS:
Overall Officials: wei wang, doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Tang ZP, Shi YH, Yin XP, Xu JZ, Zhang SM, Wang W. Modifying the details of aspiration operation may contribute to the improvement of prognosis of patients with ICH. Turk Neurosurg. 2012;22(1):13-20. doi: 10.5137/1019-5149.JTN.4219-11.0. PMID 22274965